CLINICAL TRIAL: NCT06057922
Title: A Multicenter, Open-Label, Phase 1/2 Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Patients With Selected Advanced Solid Tumors
Brief Title: A Study YL201 in Patients With Selected Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-101-01
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
Keywords: Antibody-drug conjugate
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 dose expansion stage (Experimental): Patients will be treated with YL201 intravenous (IV) infusion once every 3 weeks (Q3W) as a cycle; and at dose levels of 1.0 mg/kg and 1.2 mg/kg administered on Days 1 and 8 of each Q3W treatment cycle.
  Interventions: Drug: YL201 for Injection
- Phase 2 stage with expanded sample size (Experimental): Patients will be treated with YL201 intravenous (IV) infusion at PR2D once every 3 weeks (Q3W) as a cycle; and at dose levels of 1.0 mg/kg and 1.2 mg/kg administered on Days 1 and 8 of each Q3W treatment cycle.
  Interventions: Drug: YL201 for Injection

INTERVENTIONS:
Drug: YL201 for Injection — Patients will be treated with YL201 intravenous (IV) infusion once every 3 weeks (Q3W) as a cycle; and at dose levels of 1.0 mg/kg and 1.2 mg/kg administered on Days 1 and 8 of each Q3W treatment cycle.

SUMMARY:
This is A Multicenter, Open-Label, Phase 1/2 Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of YL201 in Patients with Selected Advanced Solid Tumors. The study will include 2 parts: Phase 1 dose expansion stage (Part 1) followed by a Phase 2 stage with expanded sample size (Part 2).

Part 1 will estimate the RP2D in dose expansion cohorts of patients with not linited to non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), nasopharyngeal carcinoma (NPC), esophageal squamous cell carcinoma (ESCC), metastatic castration-resistant prostate cancer (mCRPC), head and neck squamous cell carcinoma (HNSCC), sarcoma, ductal adenocarcinoma of pancreas (PDAC), hepatocellular carcinoma (HCC), biliary tract cancer (BTC), etc..

Part 2 will include patients with selected advanced solid tumor types enrolled at the RP2D to further assess the efficacy and safety of YL201.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the trial before the start of the trial and voluntarily sign their name and date on the ICF.
* Age ≥18 years old and ≤75 years old
* Histologically or cytologically confirmed at diagnosis of NSCLC/SCLC/NPC/ESCC /mCRPC/HNSCC/Sarcoma/PDAC/HCC/BTC
* At least one extracranial measurable lesion according to RECIST 1.1.
* Archived or fresh tumor tissue samples can be provided.
* Eastern Cooperative Oncology Group - performance scale (ECOG PS) score of 0 or 1.
* Female subjects with fertility must agree to take high-efficiency contraceptive measures from screening to whole study period and within at least 6 months after last administration of investigational drug. Male subjects must agree to take high-efficiency contraceptive measures from screening to whole study period and within at least 6 months after last administration of investigational drug.
* Life expectancy ≥3 months.
* Capable or willing to observe the visits and procedures stipulated in study protocol.

Exclusion Criteria:

* Prior treatment with products targeting B7H3 (including antibodies, antibody-drug conjugate [ADC], chimeric antigen receptor T cells [CAR-T], and other drugs).
* Prior treatment with topoisomerase 1 inhibitors or ADC based on topoisomerase 1 inhibitors.
* Participation in another clinical trial meanwhile, except observatory (non-interventional) clinical trial or at follow-up period of interventional study.
* Washout period of previous anticancer treatment was insufficient before first administration of investigational drug.
* Major surgery (excluding diagnostic surgery) within 4 weeks before first administration of investigational drug or likely to require major surgery during the study.
* History of allogenic bone marrow transplantation or solid organ transplantation.
* Treatment with systemic steroid (Prednisone >10 mg/d or equivalent drugs) or other immunosuppressive drugs within 2 weeks before first administration of investigational drug.
* Live vaccination within 4 weeks before first administration of investigational drug or likely to require live vaccine inoculation during the study.
* Evidence of leptomeningeal metastasis or carcinomatous meningitis.
* Evidence of brain metastasis or spinal cord compression.
* Evidence of cardiovascular disease with uncontrolled state or clinical significance.
* Clinically significant concomitant lung disease.
* Diagnosed as Gilbert syndrome.
* Complicated with uncontrolled third-space effusion .
* History of gastrointestinal perforation and/or fistula within 6 months before first administration.
* History of serious infection (Grade ≥3 of NCI CTCAE) before first administration.
* Known as infection with human immunodeficiency virus (HIV).
* Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
* History of any other primary malignant tumor within 5 years before first administration of investigational drug.
* The toxicity of previous anticancer treatment is not resolved.
* History of serious hypersensitive reactions to drug substance, inactive compositions of preparations or other monoclonal antibodies.
* Breastfeeding women. Or women confirmed as pregnant through pregnancy test within 3 days before first administration.
* Any disease, medical state, organ/system dysfunction or social state considered by investigators as possibly interfering the subject's capability for ICF signing, producing adverse influence on the subject's capability for cooperation and study participation or influencing the interpretation of study results. Including but not limited to mental disease or substance/alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the AEs as characterized by type, frequency, severity, timing, seriousness and relationship to study treatment | By the global end of trial date, approximately within 36 months
Evaluate the objective response rate (ORR) for patients with solid tumors which assessed using RECIST version 1.1 | Time Frame: Approximately within 36 months
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Evaluate the prostate-specific antigen (PSA) response rate for patients with prostate cancer | Time Frame: Approximately within 36 months
  PSA response rate: defined as the proportion of patients who achieved a ≥50% decrease in PSA from baseline

SECONDARY OUTCOMES:
Characterize the PK parameter AUC | Approximately within 36 months
Characterize the PK parameter Cmax | Approximately within 36 months
Characterize the PK parameter Ctrough | Approximately within 36 months
Characterize the PK parameter CL | Approximately within 36 months
Characterize the PK parameter Vd | Approximately within 36 months
Characterize the PK parameter t1/2 | Approximately within 36 months
Assess the incidence of anti-YL201 antibodies | Approximately within 36 months
Evaluate the disease control rate (DCR) for patients assessed using RECIST version 1.1 | DCR: defined as the proportion of patients who achieved a best overall response of CR, PR or stable disease (SD).
  Approximately within 36 months
Evaluate the duration of response (DoR) for patients assessed using RECIST version 1.1 | DoR: defined as the time interval from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of PD. DoR will be assessed for patients with a response (CR or PR) only.
  Approximately within 36 months
Evaluate the time to response (TTR) for patients assessed using RECIST version 1.1 | Approximately within 36 months
  TTR: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of objective response (CR or PR).
Evaluate the progression-free survival (PFS) for patients assessed using RECIST version 1.1 | Approximately within 36 months
  PFS: defined as the time interval from the date of the first dose of study drug to the date of first documentation of PD or death due to any cause, whichever occurs first.
Evaluate the overall survival (OS) for patients | Approximately within 36 months
  OS: defined as the time interval from the date of the first dose of study drug to the date of death due to any cause.
Evaluate the radiographic progression-free survival (rPFS) for patients with prostate cancer | Approximately within 36 months
Evaluate the time to PSA progression (TTPP) for patients with prostate cancer | Approximately within 36 months
  Defined as the time from the first investigational drug administration to the first recording of PSA progression.
Evaluate the PSA duration of response (PDoR) for patients with prostate cancer | Approximately within 36 months
  Defined as the time from PSA reduction of ≥50% compared with baseline to PSA progression.
Evaluate the best PSA response for patients with prostate cancer | Approximately within 36 months
  Defined as the maximum percentage of PSA changes at any time during the study.

CONTACTS AND LOCATIONS:
Locations (56):
- China (56):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The Frist People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Jiangyin People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Jiangxi Cancer Hospital (Jiangxi Second People's Hospital), Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The Frist Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanxi Cancer Hospital, Datong, Shanxi
  - The Second Affiliated Hospital of the Chinese People's Liberation Army Air Force Medical University, Xian, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Huaxi, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

REFERENCES:
- [Derived] Ma Y, Yang Y, Huang Y, Fang W, Xue J, Meng X, Fan Y, Fu S, Wu L, Zheng Y, Liu J, Liu Z, Zhuang W, Rosen S, Qu S, Li B, Li M, Zhao Y, Yang S, Ji Y, Sommerhalder D, Luo S, Yang K, Li J, Lv D, Zhang P, Zhao Y, Hong S, Zhang Y, Zhao S, Chin S, Zhang X, Lian W, Cai J, Xue T, Zhang L, Zhao H. A B7H3-targeting antibody-drug conjugate in advanced solid tumors: a phase 1/1b trial. Nat Med. 2025 Jun;31(6):1949-1957. doi: 10.1038/s41591-025-03600-2. Epub 2025 Mar 13. PMID 40082695